CLINICAL TRIAL: NCT00858169
Title: Taichung Veterans General Hospital
Brief Title: Assessment of Wrist Joint and Knee Joint Inflammation in Patients With Rheumatoid Arthritis by Quantitative Three Dimensional Power Doppler Ultrasonography
Acronym: 3D sono in RA
Status: Completed | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, TCVGH, Taichung Veterans General Hospital, Taichung Veterans General Hospital
Other Study IDs: C09044
Record Dates: First submitted 2009-03-06; First posted 2009-03-09 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Rheumatoid Arthritis
Keywords: three-dimensional power Doppler ultrasonography; wrist; knee; rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to:

1. To investigate the wrist joint synovial blood flow intensity and model by quantitative three-dimensional (3D) power Doppler ultrasonography (PDUS) in patients with rheumatoid arthritis before and after initiation of a new medicine and compare these data with routinely used clinical data and laboratory findings, such as pain score, erythrocyte sedimentation rate (ESR) and C-reactive protein (CRP)
2. To investigate the intra-observer and inter-observer agreement of quantitative 3D PDUS assessment of the vascularity in wrist joints and knee joints using automatic volume scan.

ELIGIBILITY:
Inclusion Criteria:

* Patients who fulfill the 1987 ARA criteria for RA
* Patients with at least one painful swollen wrist or knee joint observed by a rheumatologist
* Patients who will receive a new medicine, including oral corticosteroid, intravenous methylprednisolone pulse therapy, intraarticular injection with steroid or methotrexate, DMARDs, or biologic agent

Exclusion Criteria:

* Patients with active infection
* Patients with concurrent malignant disease
* Patients with a history of traumatic, septic, or cystal arthritis, previous joint surgery, or arthroscopic synovectomy of any wrist or kneejoint within the past 12 months before the study
* Patients who have severe wrist or knee joint deformity that makes the US assessment protocol unable to complete

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 30 patients with RA who visit outpatient clinic of Rheumatology at Taichung Veterans General Hospital (TCVGH) will be enrolled consecutively at if they met the study inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2009-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Correlation between 2D- and 3D-PDUS quantification data and clinical data, including pain score, erythrocyte sedimentation rate (ESR) and C-reactive protein (CRP) | cross-sectional